CLINICAL TRIAL: NCT05495152
Title: Adjuvant Sintilimab for Locally Advanced Esophageal Squamous Cell Carcinoma: a Multi-Centre, Open-Label, Randomized, Controlled, Clinical Trial (HCHTOG2203)
Brief Title: Adjuvant Sintilimab for Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Haibo Sun, Vice Chief, Department of Thoracic Surgery, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCHTOG2203
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjuvant Arm (Experimental): Patients in arm A receive 17 cycles of Sintilimab within 4 to 12 weeks after esophagectomy for ESCC. Sintilimab was administered intravenously at a dose of 200 mg over 30 minutes every 3 weeks.
  Interventions: Drug: Sintilimab
- Observation Arm (No Intervention): Patients in observation arm receive routine follow-up after surgery.

INTERVENTIONS:
Drug: Sintilimab — Patients in adjuvant arm receive 17 cycles of Sintilimab within 4 to 12 weeks after esophagectomy for ESCC. Sintilimab was administered intravenously at a dose of 200 mg over 30 minutes every 3 weeks.
  Arms: Adjuvant Arm

SUMMARY:
No adjuvant treatment has been established for patients who remain at high risk for recurrence after neoadjuvant chemotherapy plus surgery and incidental pathologic lymph node metastasis following initial surgery for esophageal squamous cell carcinoma (ESCC).Controversy still exists regarding the role of adjuvant immunotherapy for ESCC patients who do not achieve pCR after neoadjuvant chemotherapy plus surgery and clinical T1-2 N0 patients with incidental pathologic lymph node metastasis following initial surgery. To investigate the outcomes of adjuvant Sintilimab in patients with locally advanced ESCC, we initiated this randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven squamous cell carcinoma.
2. Tumours are located in the thoracic oesophagus.
3. Age is between 18 years and 70 years.
4. ECOG performance status of 0 or 1.
5. Patients with resectable cT1-4aN+M0 or T3-4aN0M0 disease and residue disease is found after neoadjuvant chemotherapy plus surgery or cT1-2N0M0 and pathologically proven T1-2N+M0 after upfront surgery.
6. No metastatic cervical lymph nodes.
7. R0 resection is achieved by the minimally invasive esophagectomy (MIE) or open McKeown approach with total two-field lymph nodes dissection or three-field lymph nodes dissection.
8. No prior therapy was administered against other cancers.
9. Adequate bone marrow function: white blood cell count ≥ 4×109/L; absolute neutrophil count (ANC) ≥ 1.5×109/l; platelets ≥ 100×109/L; haemoglobin ≥ 9 g/dl.
10. Adequate liver function: serum bilirubin ≤ 1.5 × upper limit of normal (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.0 × ULN (ULN as per institutional standard).
11. Adequate renal function: glomerular filtration rate ≥ 60 ml/min calculated using the Cockcroft-Gault formula.
12. Normal thyroid function.
13. Written consent is obtained.

Exclusion Criteria:

1. Patients receive neoadjuvant chemoradiation therapy.
2. Patients with pathological complete response (pCR).
3. No. of lymph node dissection < 15.
4. Patients with clinical stages T1-2N+M0 and receive upfront surgery.
5. Patients with unresectable disease (bulky metastatic lymph nodes or T4b) and receive induction chemotherapy.
6. Patients requiring systemic steroid medication.
7. Patients with severe postoperative complications and not suitable for adjuvant therapy.
8. Synchronous or metachronous (within 5 years) double cancers.
9. Patients ever received immunotherapy.
10. Active infection requiring systemic therapy.
11. Patients ever received organ transplant or allogenic haemopoietic stem cell transplantation.
12. Patients with human immunodeficiency virus (HIV) infection.
13. Psychiatric disease.
14. Pregnant or lactating women or women of childbearing potential.
15. Hypersensitivity for Sintilimab.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival (DFS) | DFS is defined as the time from the date of randomization to the date of first recurrence (local, regional or distant) or death , assessed up to 36 months
  DFS is defined as the time from the date of randomization to the date of first recurrence (local, regional or distant) or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Batran SE, Koch C. Neoadjuvant therapy for oesophageal cancer: refining the armamentarium. Lancet. 2024 Jul 6;404(10447):5-7. doi: 10.1016/S0140-6736(24)01084-5. Epub 2024 Jun 11. No abstract available. PMID 38876135
- [Derived] Sun HB, Xing WQ, Liu XB, Yang SJ, Chen PN, Liu SL, Li P, Ma YX, Jiang D, Yan S. A multicenter randomized, controlled clinical trial of adjuvant sintilimab for esophageal squamous cell carcinoma. Future Oncol. 2023 Aug;19(26):1777-1784. doi: 10.2217/fon-2022-1255. Epub 2023 Sep 22. PMID 37737025